CLINICAL TRIAL: NCT07371793
Title: A Phase 1/2a, Two-Part, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate Safety, Tolerability and Pharmacodynamics of Multiple Doses of Oral BBI-001 in Healthy Participants and in Participants With Hereditary Hemochromatosis
Brief Title: A Study to Evaluate BBI-001 in Healthy Volunteers and in Patients With Hereditary Hemochromatosis
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bond Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BBI-001-102
Record Dates: First submitted 2026-01-20; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Hereditary Hemochromatosis
MeSH Terms: conditions — Hemochromatosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BBI-001 (Experimental)
  Interventions: Drug: BBI-001
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: BBI-001 — In Part 1 BBI-001 administered TID for 14 days. In Part 2 BBI-001 administered TID for 3 days in a cross-over fashion.
  Arms: BBI-001
Other: Placebo — In Part 1 placebo administered TID for 14 days. In Part 2 placebo administered TID for 3 days in a cross-over fashion.
  Arms: Placebo

SUMMARY:
This study will be conducted in two parts run in parallel.

Part 1 of the study (Phase 1, randomized, double-blind, placebo-controlled, multiple ascending dose) will enroll healthy volunteers in 3 sequential dose escalating cohorts with BBI-101 or placebo administered 3 times per day (TID) for 14 days.

Part 2 of the study (Phase 2a, randomized, multiple dose, two-period, two-sequence crossover) will evaluate the effect of BBI-001 on blood iron parameters in patients with hereditary hemochromatosis receiving 8 doses of BBI-001 or placebo treatment administered TID in Period 1 followed by administration of reverse treatment in Period 2. Dosing periods will be separated by 12 days.

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers (Part 1) or patients with hereditary hemochromatosis (Part 2)

Exclusion Criteria:

Serious or unstable medical or psychiatric conditions

Significant medical history

Current infections

Alcohol use disorder

Receiving iron chelation therapy or treatment other than stable maintenance phlebotomy for the prior 6 months (Part 2)

Organ damage from iron overload in the view of the principal investigator would prevent successful completion of the protocol (Part 2)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AE) | Up to 30 days
  Incidence and severity of AEs and serious AEs (SAEs), including clinically significant abnormalities in physical examinations, vitals signs, ECG parameters, and laboratory results

CONTACTS AND LOCATIONS:
Overall Officials: Curtis Scribner, MD, Study Chair — Bond Biosciences
Locations (1):
- Clinical Research Unit, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsor website — https://bond.bio